CLINICAL TRIAL: NCT05701124
Title: Intravitreal Ranibizumab Injection In Aggressive Retinopathy Of Prematurity Compared With Type 1 Prethreshold Retinopathy Of Prematurity
Brief Title: Intravitreal Ranibizumab Injection for Aggressive Versus Type 1 Prethreshold Retinopathy of Prematurity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Ghada Mahmoud Tawfik Ibrahim Eladawy, principal investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZU-IRB#6269/22-7-2020
Record Dates: First submitted 2023-01-08; First posted 2023-01-27 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Retina Disease; Retinopathy of Prematurity; Ranibizumab
Keywords: Aggressive ROP; Ranibizumab; Type 1 ROP; anti-VEGF; Laser photocoagulation
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant
Masking Description: single masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Aggressive ROP (Active Comparator): Intravitreal injection (IVI) was performed under topical anesthesia in standard ophthalmic operating room. 5% povidone-iodine disinfection and topical antibiotic were instilled. Ranibizumab (0.25 mg/0.025 mL) was injected into the vitreous cavity with a 31-gauge needle, aiming the needle directly toward the optic nerve in direction of visual axis 1.0 mm posterior to the corneoscleral junction at the inferotemporal quadrant.
  Interventions: Drug: Ranibizumab (0.25 mg/0.025 mL)
- Type 1 prethreshold ROP (Active Comparator): Intravitreal injection (IVI) was performed under topical anesthesia in standard ophthalmic operating room. 5% povidone-iodine disinfection and topical antibiotic were instilled. Ranibizumab (0.25 mg/0.025 mL) was injected into the vitreous cavity with a 31-gauge needle, aiming the needle directly toward the optic nerve in direction of visual axis 1.0 mm posterior to the corneoscleral junction at the inferotemporal quadrant.
  Interventions: Drug: Ranibizumab (0.25 mg/0.025 mL)

INTERVENTIONS:
Drug: Ranibizumab (0.25 mg/0.025 mL) — Intravitreal injection (IVI) was performed under topical anesthesia in standard ophthalmic operating room. 5% povidone-iodine disinfection and topical antibiotic were instilled. Ranibizumab (0.25 mg/0.025 mL) was injected into the vitreous cavity with a 31-gauge needle, aiming the needle directly toward the optic nerve in direction of visual axis 1.0 mm posterior to the corneoscleral junction at the inferotemporal quadrant. The intraocular pressure and central artery perfusion were then checked.
  Other Names: Lucentis

SUMMARY:
Despite advances in the neonatal intensive care units, retinopathy of prematurity (ROP) has become a common reason for blindness and visual disabilities in premature infants so that it accounts for about 5% and 30% of such complications in developed and developing countries. The pathophysiology of ROP is multifactorial. Supplemental oxygen demand and lower gestational age (GA) and birth weight (BW) are among the major risk factors for the occurrence and progression of ROP.

Anti-vascular endothelial growth factor (anti-VEGF) agents are a promising modality of treatment for ROP, as laser therapy is associated with disadvantages such as complications from undertreatment or overtreatment, anterior segment burns, hemorrhage, or ischemia, and potentially higher rates of myopia. Ranibizumab is the first approved anti-VEGF treatment for the management of retinopathy, and is a promising alternative to laser therapy.

Ranibizumab is a humanized monoclonal recombinant antibody fragment with a shorter half-life and less systemic toxicity than bevacizumab. Its binding affinity is nearly tenfold that of bevacizumab.

The plasma half-life of bevacizumab is 17-21 days, while that of ranibizumab is 3 days. Greater systemic absorption of bevacizumab is thought to lead to greater systemic suppression of VEGF. These data may explain the better safety profile of ranibizumab. Type I ROP is defined as any stage of ROP with plus disease in zone I, stage 3 ROP in zone I and stage 2 or 3 ROP with plus disease in zone II . The hallmark of Aggressive-ROP (previously known as Aggressive posterior-ROP) is rapid development of pathological neovascularization and severe plus disease without progression being observed through the typical stages of ROP. It may occur in larger preterm infants and beyond the posterior retina.

The aim of this prospective study is to compare the efficacy of intravitreal ranibizumab for type 1 ROP and A-ROP as regard acute ROP regression, recurrence profile, peripheral retinal vascularization and the need for further ablative therapy.

DETAILED DESCRIPTION:
A prospective randomized study of 37 eyes of 30 infants, who received intravitreal injections of ranibizumab in one eye (the most severe) or both eyes, were included. A-ROP group included 18 eyes of 15 infants and type 1 ROP group included 19 eyes of 15 infants. The primary outcome measure was the number of eyes that achieved regression of ROP without additional treatment till 55 weeks' post-menstrual age (PMA). The mean follow-up period for A-ROP group was 11.44 months and 13.95 months for type 1 ROP group.

Treatment was performed within 72 hours once treatment criteria were detected. Intravitreal injection (IVI) was performed under topical anesthesia in standard ophthalmic operating room. 5% povidone-iodine disinfection and topical antibiotic were instilled. Ranibizumab (0.25 mg/0.025 mL) was injected into the vitreous cavity with a 31-gauge needle, aiming the needle directly toward the optic nerve in direction of visual axis 1.0 mm posterior to the corneoscleral junction at the inferotemporal quadrant. The intraocular pressure and central artery perfusion were then checked. Topical antibiotics were given for 7 days postoperatively. All infants were followed up on the next day, third day, then weekly until the regression of ROP, after that every (2-4) weeks until a minimum of 55 weeks' post menstrual age (PMA) or retinal vascularization achieved zone III without an active component such as hemorrhage or exudation or clinically significant tractional elements, which came earlier. Each examination evaluated disease regression (via indirect fundoscopic analysis), recurrence, the presence of tractional elements and peripheral vascularization. Then follow up was continued monthly for at least 6 months following treatment.

Successful treatment was defined as remission of plus disease, good pupil dilation and reduced disease grade. Outcomes were further classified as insufficient regression (persistence of plus disease and neovascularization at 3-5 days' post-injection), progression (post-injection intravitreal hemorrhage, increased neovascularization and formation of tractional components) and recurrence requiring treatment (recurrence of plus disease, recurrent neovascularization, reformation of a ridge or extraretinal fibrovascular proliferation, despite initial regression post injection) Once insufficient regression or ROP recurrence requiring treatment was determined, rescue therapy of IVR was applied.

Cases with no recurrence or recurrence not requiring treatment (stage 1 or 2 eyes, with Zone 2 or Zone 3 localisation, not accompanied by plus disease) were closely monitored until peripheral retinal vascularization was completed.

In case of failed peripheral retinal vascularization to approach zone III until 55 weeks' PMA, an indirect infrared diode laser (IRIDEX, Iris Medical SL laser with laser indirect ophthalmoscope (LIO) Ophthalmic Laser, 810 nm, USA) was used to apply photocoagulation through a +20/+28 diopter condensing lens under sedation or general anesthesia in the operating room to reduce the risk of late ROP reactivation.

Follow-up examinations were made weekly for the first month after laser photocoagulation and at 3-4-week intervals thereafter until the ROP findings receded. Follow-up examinations were continued at 3-4-month intervals after the patients turned 1-year old.

ELIGIBILITY:
Inclusion Criteria:

* Infants with a birth weight of ≤ 1500 g or gestational age of ≤ 30 weeks and selected infants with birth weight between 1500 and 2000 g or gestational age of more than 30 weeks with an unstable clinical course, including those requiring cardiorespiratory support.
* Infants with type 1 ROP, as defined by the ETROP study 11, Zone 1, any stage ROP with plus disease; Zone 1, stage 3 ROP with or without plus disease; Zone 2, stage 2 or 3 ROP with plus disease( affecting either one or both eyes).
* Aggressive ROP (A-ROP), according to the International Classification of ROP (ICROP) criteria affecting either one or both eyes.

Exclusion Criteria:

* Eyes with previous intravitreal injections.
* Eyes with previous laser therapy.
* Eyes with any other pathology, other than ROP.
* Eyes with ROP stage 4 or 5.

Ages: 28 Days to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2022-11-20 (Actual)

PRIMARY OUTCOMES:
Number of eyes that achieved regression of plus disease or active neovessels achieved either by single or multiple injections | at 55 weeks post-menstrual age
  active ROP regression
The number of eyes in which retinal vessels reach ora serrata (complete retinal vascularization) | at 55 weeks post-menstrual age
  complete retinal vascularization(retinal vessels reach ora serrata)

SECONDARY OUTCOMES:
The number of eyes that showed recurrent plus disease, recurrent neovascularization, reformation of a ridge | at 55 weeks post-menstrual age
  Recurrence requiring retreatment
The number of eyes that needed late peripheral laser | at 55 weeks post-menstrual age
  avascular peripheral retina that needed laser
The number of eyes progressing to stage 4 or 5 necessitating vitrectomy with/without lensectomy | one year
  retinal detachment(stage 4 or 5)

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Abbas Dabour, MD, FRCS, Study Director — Zagazig University
Locations (1):
- Zagazig University, Faculty of medicine, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No